CLINICAL TRIAL: NCT02077829
Title: Implementation of Illness Management and Recovery in Mental Health Services: Facilitators and Barriers in the Implementation Process.
Brief Title: Implementation of Illness Management and Recovery in Mental Health Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: Romeriksprosjektet (Unknown); Helse Sor-Ost (Other Government)
Responsible Party: Principal Investigator, Kristin Sverdvik Heiervang, Researcher, University Hospital, Akershus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IMR 01/2014; 2013/2035b (Registry Identifier: Reginal Ethical Committee)
Record Dates: First submitted 2014-02-25; First posted 2014-03-04 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Bipolar Disorder; Schizophrenia; Affective Disorders, Psychotic; Mood Disorders; Mental Disorders
Keywords: Implementation process; implementation strategy; Implementation research; evidence based practice; recovery; Illness management and recovery
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia; Affective Disorders, Psychotic; Mood Disorders; Mental Disorders | interventions — Salvage Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMR therapists, IMR patients (Other): 30 voluntary therapists from 9 mental health services will be trained and coached in IMR.
  40 patients from the 9 mental health services will receive Illness Management and Recovery from the therapists in training.
  Interventions: Behavioral: Illness Management and Recovery

INTERVENTIONS:
Behavioral: Illness Management and Recovery — Evidence-based practice given individually or in groups, weekly for 10-12 months.
  Other Names: IMR

SUMMARY:
The purpose of this study is to examine the barriers and facilitators of implementing Illness Management and Recovery (IMR) in Norwegian mental health services.

DETAILED DESCRIPTION:
IMR is an evidence-based practice developed for people with severe mental illnesses. It is based on the principles of recovery to help people set individual meaningful goals for their lives and gain illness self-management skills and thereby contribute to their individual recovery-process. IMR can be given individually or in groups, once a week for 10-12 months.

In this project the investigators will implement Illness Management and Recovery (IMR) in mental health services. The implementation strategy are carried out according to the IMR toolkits which include informational and training materials, implementation recommendations, and fidelity scales to facilitate use of the model in routine practices. The implementation process and outcome will be of main focus.

The study has an observational prospective cohort design. 30 therapists from 9 different mental health services will be trained and supervised in IMR. The investigators aim to enrol 40 patients. The primary outcome is therapists' fidelity to the model and organisational implementation outcome. Secondary outcomes are patients' level of functioning and hope.

ELIGIBILITY:
Inclusion Criteria Therapists:

* Voluntary recruited therapists in the participating mental health services
* trained and consulted in IMR

Inclusion Criteria Patients:

* Adults (18+)
* Associated with one of the participating mental health services
* symptoms on or diagnosis of severe mental illness with or without drug abuse
* giving informed consent verbally and in writing

Exclusion Criteria Patients:

* Patients with acute risk of suicidal behaviour
* not able to communicate in Norwegian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The Illness Management Fidelity Scale (SAMHSA, 2009) | 12 months
  Assesses the degree of fidelity with 13 items on a 5-point likert scale where 5 indicates full implementation and 0 indicates no implementation

SECONDARY OUTCOMES:
The Illness Management & Recovery Treatment Integrity Scale (IT-IS) (McGuire et al., 2012 | 12 months
  A 16-item scale measuring clinicians' faithful replication of the model
The Adult State Hope Scale (Snyder et al., 1996) | 12 months
  A 6-item self-report scale of patients' hope and optimism
The Illness Management and Recovery Scale (SAMHSA, 2009) | About 11 months after start of intervention
  Assessing patients' recovery outcomes in the IMR program with 15 items.
General Organizational Index (SAMHSA, 2009) | 12 months
  A 12-item scale measuring organisational outcome of implementation by common agency practices that support evidence-based practices

CONTACTS AND LOCATIONS:
Overall Officials: Kristin S. Heiervang, Ph.D., Principal Investigator — Akershus University Hospital, Research & Development, Mental Health Services
Locations (1):
- Ahus R&D Mental Health Services, Lørenskog, Norway

REFERENCES:
- [Derived] Egeland KM, Hauge MI, Ruud T, Ogden T, Heiervang KS. Significance of Leaders for Sustained Use of Evidence-Based Practices: A Qualitative Focus-Group Study with Mental Health Practitioners. Community Ment Health J. 2019 Nov;55(8):1344-1353. doi: 10.1007/s10597-019-00430-8. Epub 2019 Jun 12. PMID 31190179
- [Derived] Egeland KM, Ruud T, Ogden T, Fardig R, Lindstrom JC, Heiervang KS. How to implement Illness Management and Recovery (IMR) in mental health service settings: evaluation of the implementation strategy. Int J Ment Health Syst. 2017 Jan 23;11:13. doi: 10.1186/s13033-017-0120-z. eCollection 2017. PMID 28127388